CLINICAL TRIAL: NCT01009931
Title: A Phase II Study of 12-O-tetradecanoylphorbol-13-acetate (TPA) Plus Dexamethasone & Choline Magnesium Trisalicylate in the Treatment of Patients With Relapsed/Refractory Acute Myelogenous Leukemia
Brief Title: Phase II Study of TPA Plus Dexamethasone & CMT in Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to lack of experimental medication (supply issues)
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH); Biosuccess Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020702; P30CA068485 (NIH); 0220080085 (Other: IRB #); P30CA072720 (NIH); NCI-2011-03242 (Other: CTRP (Clinical Trails Reporting Program))
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Tetradecanoylphorbol Acetate; Dexamethasone; dexamethasone 21-phosphate; choline magnesium trisalicylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPA + Dexamethasone and CMT (Experimental): 12-O-tetradecanoylphorbol-13-acetate (TPA) plus Dexamethasone & Choline magnesium trisalicylate (Trilisate)
  Interventions: Drug: 12-O-tetradecanoylphorbol-13-acetate; Drug: Dexamethasone; Drug: Choline magnesium trisalicylate

INTERVENTIONS:
Drug: 12-O-tetradecanoylphorbol-13-acetate — The initial dose of TPA will be 1 mg/week x 3 weeks (Day 1, 8, 15). Up to 6 cycles.
  Other Names: TPA
Drug: Dexamethasone — Dexamethasone 10 mg PO qid will start 24h prior to TPA and continue for 24h after TPA x 3 weeks. Up to 6 cycles.
  Other Names: Dexamethasone sodium phosphate
Drug: Choline magnesium trisalicylate — Choline magnesium trisalicylate 1500 mg PO TID will begin 24h prior to TPA and continue for 24h post TPA x 3 weeks.
  Up to 6 cycles.
  Other Names: Trilisate

SUMMARY:
This phase II trial is studying the side effects and how well giving tetradecanoylphorbol acetate together with dexamethasone and choline magnesium trisalicylate works in treating patients with relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria

* Must have a histologically documented relapsed/refractory AML for which there is no standard therapy that has been demonstrated to have curative or palliative potential.
* ECOG performance status of 0-2.
* Must be 18 years or older.
* Estimated life expectancy > 1 month.
* Laboratory data:

  * total bilirubin ≤ 1.5 x upper limit of normal unless due to Gilbert's syndrome
  * serum creatinine ≤ 2.0 mg/dl
  * AST ≤ 3.0 x upper limit of normal
  * Cardiac ejection fraction > 40%
  * FEV1.0 > 50% predicted
* Prior therapy: > 3 weeks since chemotherapy, biological therapy or radiation; anticipated maximum hematological improvement since last dose of chemotherapy. (Concurrent hydroxyurea administration will be allowed to control WBC count, platelet count, or symptoms).
* No active infections.
* Negative pregnancy test for women of childbearing potential.
* No uncontrolled psychiatric illness or medical illness that the principal investigator feels will compromise the patient's tolerance of the study medication.
* Must provide informed consent.

Exclusion Criteria

* Patients with an allergy to proton pump inhibitors, required for GI prophylaxis; or salicylates are excluded.
* Pregnant or lactating women
* Age <18 years. Because no dosing or adverse event data are currently available on the use of TPA alone or in combination with dexamethasone in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric Phase II combination trials.
* The effects of TPA on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 10 weeks after. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Should the female partner of a participant in this study become pregnant or suspect she is pregnant during this study, the PI of this study will be available to provide advice about further medical/obstetric care/referral for the female partner.
* Patients with active CNS involvement (documented by radiographic lesions and/or malignant cells in the CSF) will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with treatment of any other investigational drug within the last 30 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TPA + Dexamethasone and CMT: 12-O-tetradecanoylphorbol-13-acetate (TPA) plus Dexamethasone & Choline magnesium trisalicylate (Trilisate)
  12-O-tetradecanoylphorbol-13-acetate: The initial dose of TPA will be 1 mg/week x 3 weeks (Day 1, 8, 15).
  Up to 6 cycles.
  Dexamethasone: Dexamethasone 10 mg PO qid will start 24h prior to TPA and continue for 24h after TPA x 3 weeks. Up to 6 cycles.
  Choline magnesium trisalicylate: Choline magnesium trisalicylate 1500 mg PO TID will begin 24h prior to TPA and continue for 24h post TPA x 3 weeks.
  Up to 6 cycles.
Period: Overall Study
Arm/Group | TPA + Dexamethasone and CMT
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPA + Dexamethasone and CMT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate > 20% for 12-O-tetradecanoylphorbol-13- Acetate (TPA)+ Dexamethasone + Choline Magnesium Trisalicylate(Trilisate)
Time Frame: 42 months
Population: The study participant died before the study data collection completed.
Arm/Group | TPA + Dexamethasone and CMT
Number analyzed (Participants) | 0

2. Primary Outcome: Grade 3 and 4 Non-hematologic Treatment-related Toxicity Rates < 25%
Time Frame: 43 months
Population: The study participant died before the study data collection completed.
Arm/Group | TPA + Dexamethasone and CMT
Number analyzed (Participants) | 0

3. Secondary Outcome: Effects of Treatment on Immunophenotype, Signaling Profile, and Nuclear NF-kB Expression
Description: Cycle 1 of treatment
Time Frame: 48 months
Population: The study participant died before the study data collection completed.
Arm/Group | TPA + Dexamethasone and CMT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | TPA + Dexamethasone and CMT
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPA + Dexamethasone and CMT (N=1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 1 (2)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes